CLINICAL TRIAL: NCT07254026
Title: Developing a Precision Health Approach for Obstructive Sleep Apnea: Treatment Responses Analysis and Smart Telerehabilitation Systems
Brief Title: Precision Health and Smart Telerehabilitation in OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-114-020
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surgical Procedures, Operative; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Surgical (Experimental): Surgery for OSA
  Interventions: Procedure: Surgery
- Continuous positive airway pressure (Experimental): Receive continuous positive airway pressure
  Interventions: Device: Continuous positive airway pressure
- Oropharyngeal rehabilitation with diary (Experimental): Receive oropharyngeal telerehabilitation training over three months
  Interventions: Other: Oropharyngeal Exercise with diary
- Oropharyngeal rehabilitation with smartphone application (Experimental): Receive oropharyngeal telerehabilitation training incorporated with a smartphone application (Adaptive Sensor-Based Motion Tracking, ASMT system, which consisted of a pressure sensor and facial motion recognition technology) for over three months
  Interventions: Other: Oropharyngeal Exercise with smartphone application

INTERVENTIONS:
Procedure: Surgery — Including septomeatoplasty, uvulopalatopharyngoplasty (UPPP), or/and tongue base reduction surgery.
  Arms: Surgical
Device: Continuous positive airway pressure — Continuous positive airway pressure, 1-5 days a week for three months.
  Arms: Continuous positive airway pressure
Other: Oropharyngeal Exercise with diary — Oropharyngeal exercise conducted via the telerehabilitation method. Participants are required to attend online supervised sessions of exercises 1-5 days a week for three months. Participants are required to fill out the exercise diary upon completion of the training each day.
  Arms: Oropharyngeal rehabilitation with diary
Other: Oropharyngeal Exercise with smartphone application — Oropharyngeal exercise conducted via the telerehabilitation method. Participants are required to attend online supervised sessions of exercises 1-5 days a week for three months. In addition to attending the weekly supervised telerehabilitation sessions online, these participants will independently perform the exercises using the smartphone application incorporated with ASMT one to three times per week, with each session lasting approximately 45-60 minutes.
  Arms: Oropharyngeal rehabilitation with smartphone application

SUMMARY:
This study aims to improve treatment strategies for Obstructive Sleep Apnea (OSA), a disorder characterized by recurrent upper airway collapse during sleep, resulting in reduced oxygenation, sleep fragmentation, and excessive daytime sleepiness. The objectives are twofold: to evaluate whether an artificial intelligence (AI)-based model can accurately predict the most effective treatment for individual patients, and to assess whether a mobile health application can enhance adherence to oropharyngeal rehabilitation (OPR) and improve therapeutic outcomes.

The study will be conducted in two phases. In Phase I, a retrospective analysis will be performed using a large dataset of polysomnography (PSG) records obtained from the Sleep Center at National Cheng Kung University Hospital. Machine learning algorithms will be applied to identify predictive features that differentiate responders from non-responders across Continuous Positive Airway Pressure (CPAP), surgical, and OPR interventions. These findings will inform the development of a predictive treatment recommendation model.

In Phase II, a prospective clinical trial will validate the predictive accuracy and clinical utility of the model. Patients newly diagnosed with OSA will be assigned to CPAP, surgery, or OPR interventions according to the model's recommendations, in combination with physician judgment and patient preference. Each intervention will last 12 weeks, followed by repeat PSG and clinical assessments. Within the OPR arm, participants will be further randomized to monitor adherence via an exercise diary or a smartphone application equipped with a pressure sensor and facial motion recognition technology, enabling real-time feedback and remote monitoring.

This trial is expected to determine whether AI can provide clinically reliable treatment recommendations and whether digital telerehabilitation can improve adherence and outcomes, thereby advancing precision medicine in OSA management.

DETAILED DESCRIPTION:
This study is designed to improve treatment strategies for Obstructive Sleep Apnea (OSA), a disorder characterized by reduced oxygenation and recurrent sleep disturbances. The research has two primary objectives: first, to evaluate whether an artificial intelligence (AI)-based model can accurately predict the most effective treatment for individual patients; and second, to assess whether a mobile health application can facilitate oropharyngeal exercise training, thereby enhancing adherence and therapeutic outcomes.

The study will be conducted in two phases. In Phase I, researchers will analyze a large dataset of polysomnography (PSG) records obtained from the Sleep Center at National Cheng Kung University Hospital. Machine learning methods will be applied to identify predictive patterns that distinguish responders from non-responders across treatments such as Continuous Positive Airway Pressure (CPAP), surgical intervention, and oropharyngeal rehabilitation (OPR).

In Phase II, a prospective clinical trial will be implemented. Patients newly diagnosed with OSA will be allocated to CPAP, surgical, or OPR interventions (with either an exercise diary or a smartphone application) according to the AI-generated treatment recommendations, supplemented by physician judgment and patient preference. Each intervention will last 12 weeks, after which repeat PSG and clinical evaluations will be conducted to assess treatment efficacy.

Participants in the CPAP arm will undergo 12 weeks of nightly CPAP use. Participants in the surgical group will receive operative treatment for OSA. Those assigned to the OPR arm will complete 12 weeks of telerehabilitation training focused on oropharyngeal exercises. Within the OPR group, participants will be further divided into two subgroups: one will record adherence using an exercise diary, while the other will train with a smartphone application integrated with a pressure sensor and facial motion recognition technology. This system will provide real-time feedback, record adherence, and transmit performance data to a secure cloud platform, enabling remote monitoring and clinician-guided adjustments.

The study aims to determine whether AI can deliver clinically reliable, personalized treatment recommendations and whether app-based telerehabilitation can improve adherence and treatment outcomes. The anticipated results are expected to advance precision medicine approaches in OSA management and enhance both patient care and healthcare efficiency.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old and above
* Newly diagnosed with mild to severe pure obstructive sleep apnea based on polysomnography

Exclusion Criteria:

* Severe allergic rhinitis
* Sinusitis with nasal polyps
* Body Mass Index (BMI) > 31
* Alcohol or drug abuse within the past year
* Pregnancy
* Severe obstructive or restrictive pulmonary diseases
* High-risk cardiovascular diseases during exercise (e.g., angina, myocardial infarction, heart failure, valvular heart disease)
* History of central or peripheral neurological disorders that interfere with exercise prescription
* Musculoskeletal or psychological disorders that interfere with exercise prescription
* Other non-respiratory sleep disorders
* Sleep disorders with concomitant central sleep apnea

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | Baseline and 12 weeks post intervention
  The apnea-hypopnea index will be obtained from the overnight Polysomnography (PSG) study. PSG will be performed in the sleep center of National Cheng Kung University Hospital. Less than 5 events/hour indicates normal; AHI between 5-14 events/hour indicates mild Obstructive Sleep Apnea(OSA); AHI between 15-30 events/hour indicates moderate OSA; and AHI more than 30 events/hour indicates severe OSA.

SECONDARY OUTCOMES:
Daytime Sleepiness Level | Baseline and 12 weeks post intervention
  Epworth Sleepiness Score(ESS) will be used to measure the daytime sleepiness of OSA patients. The total score of ESS range from 0-24. A score greater than 10 indicates greater daytime sleepiness.
Sleep Quality | Baseline and 12 weeks post intervention
  Sleep quality will be measured using Pittsburgh Sleep Quality Index (PSQI).The total score ranges from 0 to 21 with a higher total score equal to or more than 5 indicating worse sleep quality.
Pharyngeal Airway Volume | Baseline and 12 weeks post intervention
  Computer Tomography (CT) will be performed. The pharyngeal airway volume will be calculated from the hard palate to the epiglottis and the data will be presented in cm^3. The minimum score is 0 and a higher score indicates greater in pharyngeal airway volume.
Cross Section Area on the Tip of Epiglottis | Baseline and 12 weeks post intervention
  Computer Tomography (CT) will be performed. Cross section area on the tip of the epiglottis was measured and the data will be presented in cm^2. The minimum score is 0 and a higher score indicates greater in the cross-sectional area of the region.
Anterior to Posterior Distance on the Tip of the Epiglottis | Baseline and 12 weeks post intervention
  The distance between the anterior and posterior pharyngeal wall on the tip of the epiglottis will be measured and presented in cm. The minimal value will be 0 and the greater value indicates a greater distance between the anterior to posterior in this area.
Lateral Distance on the Tip of Epiglottis | Baseline and 12 weeks post intervention
  The distance between the lateral distance on the tip of the epiglottis will be measured and presented in cm. The minimal value will be 0 and the greater value indicates a greater distance between the lateral wall.
Median Usage Hours of Continuous Positive Airway Pressure | 1-week average pre intervention, 1-week average post intervention and 1-month average during intervention for 3 months
  The average number of hours per night that participants use CPAP will be recorded from CPAP usage reports. Greater nightly usage is considered indicative of better compliance and treatment effectiveness.
Median Pressure in Continuous Positive Airway Pressure | 1-week average pre intervention, 1-week average post intervention and 1-month average during intervention for 3 months
  The change in therapeutic CPAP pressure required to maintain airway patency will be assessed using CPAP usage reports. A reduction in required pressure is expected to indicate improved upper airway muscle tone and stability.
Tongue Muscle Strength | Baseline and 12 weeks post intervention
  The maximal muscle strength of genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (kPa)
Tongue Muscle Endurance | Baseline and 12 weeks post intervention
  The endurance of the genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (in seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No